CLINICAL TRIAL: NCT01699295
Title: Physical Activity and Academic Achievement Across the Curriculum (A+PAAC)
Acronym: A+PAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph Donnelly (Other)
Responsible Party: Sponsor-Investigator, Joseph Donnelly, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13460
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Intelligence; Obesity
Keywords: academic achievement; elementary school; physical activity; exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A+PAAC (Experimental): Lessons delivered using A+PAAC
  Interventions: Behavioral: A+PAAC
- CON (Active Comparator): Regular sedentary lessons
  Interventions: Behavioral: CON

INTERVENTIONS:
Behavioral: A+PAAC — academic lessons delivered by regular classroom teachers using moderate to vigorous physical activity (MVPA) for 20 minutes/day, 5 days/week.
  Arms: A+PAAC
Behavioral: CON — lessons taught by regular classroom teachers using traditional/regular sedentary lessons
  Arms: CON

SUMMARY:
There is currently considerable interest in both improving academic achievement (No Child Left Behind) and reducing the rates of obesity and its associated negative health consequences in elementary school students. Increased physical activity (PA) offers a potential intervention to address both issues. Evidence is available which suggests an association of PA with both academic achievement and obesity, and an association between obesity and academic achievement.

To provide increased PA while maintaining academic instruction time, we developed a program we call "Physical Activity Across the Curriculum" (PAAC) in which regular classroom teachers were trained to deliver academic lessons using moderate to vigorous physical activity (MVPA) for 20 minutes/d, 5 days/wk. This study is looking to compare academic achievement between students in elementary schools that participate in academic lessons taught through MVPA (PAAC) to students that do not (CON).

ELIGIBILITY:
Inclusion Criteria:

* Grade 2 or 3 Student at one of the randomly selected elementary schools
* Students that agree to complete assessments
* Signed parental consent form
* Signed child assent form

Exclusion Criteria:

* Students that do not agree to complete assessments

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 584 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in Academic Achievement in Elementary Students | Baseline to 3 Years
  Changes in academic achievement between students in elementary schools that participate in a program that delivers academic lessons taught through MVPA (A+PAAC) to students in elementary schools that do not receive academic lessons taught through MVPA (CON)

SECONDARY OUTCOMES:
Assessment of Cognitive Function | Baseline to 3 Years
  Changes in attentional control and academic achievement
Body Mass Index (BMI) | Baseline to 3 Years
  Change in the BMI over course of the study.
Cardiovascular (CV) Fitness and Daily Physical Activity (PA) | Baseline to 3 Years
  Changes in CV Fitness and PA and its impact on cognitive control of attention and academic achievement
Change in Attention-to-Task | Baseline to 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, EDD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Honas JJ, Willis EA, Herrmann SD, Greene JL, Washburn RA, Donnelly JE. Energy Expenditure and Intensity of Classroom Physical Activity in Elementary School Children. J Phys Act Health. 2016 Jun;13(6 Suppl 1):S53-6. doi: 10.1123/jpah.2015-0717. PMID 27392380
- [Derived] Willis EA, Ptomey LT, Szabo-Reed AN, Honas JJ, Lee J, Washburn RA, Donnelly JE. Length of moderate-to-vigorous physical activity bouts and cardio-metabolic risk factors in elementary school children. Prev Med. 2015 Apr;73:76-80. doi: 10.1016/j.ypmed.2015.01.022. Epub 2015 Jan 31. PMID 25647532
- [Derived] Hansen DM, Herrmann SD, Lambourne K, Lee J, Donnelly JE. Linear/nonlinear relations of activity and fitness with children's academic achievement. Med Sci Sports Exerc. 2014 Dec;46(12):2279-85. doi: 10.1249/MSS.0000000000000362. PMID 24781896
- [Derived] Donnelly JE, Greene JL, Gibson CA, Sullivan DK, Hansen DM, Hillman CH, Poggio J, Mayo MS, Smith BK, Lambourne K, Herrmann SD, Scudder M, Betts JL, Honas JJ, Washburn RA. Physical activity and academic achievement across the curriculum (A + PAAC): rationale and design of a 3-year, cluster-randomized trial. BMC Public Health. 2013 Apr 8;13:307. doi: 10.1186/1471-2458-13-307. PMID 23565969